CLINICAL TRIAL: NCT00351897
Title: The Efficacy of Pulsed Dye Laser in Dermatophytosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr.Nima Ostovari
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: src-ost-1358
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2008-02-20 (Estimated); Status verified 2007-07

CONDITIONS: Cutaneous Dermatophytosis; Pulsed Dye Laser
MeSH Terms: interventions — Laser Therapy

INTERVENTIONS:
Device: pulsed dye (585nm) laser therapy

SUMMARY:
The purpose of this study is to determine whether Pulsed Dye Laser therapy are effective in the treatment of Cutaneous Dermatophytosis.

DETAILED DESCRIPTION:
This study was conducted to determine the efficacy of Pulse Dye Laser in skin fungal infection, if this study showed that Laser could be effective, this would be introduced as a new treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Positive KOH Smear skin plaques

Exclusion Criteria:

* Tinea Capitis,Onychomycosis
* Pregnancy and feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
smear & culture of skin scrap

CONTACTS AND LOCATIONS:
Overall Officials: Nima Ostovari, M.D., Study Director — Shahid Beheshti University of Medical Sciences; Parviz Toossi, MD, Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Skin Research Center, Shaheed Beheshti Medical University, Tehran, Iran